CLINICAL TRIAL: NCT00739063
Title: Study of Erlotinib, Small Molecule Targeting Epidermal Growth Factor Receptor (EGFR) in Treatment of Patients w/EGFR-overexpressing 'Triple Receptor-negative' Metastatic Carcinoma of Breast That Progressed on Anthracyclines and Taxanes
Brief Title: Phase II Study of Erlotinib, an EGFR Inhibitor in Metastatic EGFR-positive 'Triple Receptor-negative' Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0613
Record Dates: First submitted 2008-08-19; First posted 2008-08-21 (Estimated); Results first posted 2012-03-15 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Carcinoma of the breast; Stage IV; Triple receptor-negative; Triple receptor-negative breast cancer; Metastatic triple receptor-negative breast cancer; Epidermal growth factor receptor; EGFR; EGFR-overexpressing; GFR inhibitor erlotinib; Erlotinib hydrochloride; Erlotinib; Tarceva; OSI-774
MeSH Terms: conditions — Breast Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tarceva daily (Experimental): Tarceva oral 150 mg daily.
  Interventions: Drug: Tarceva

INTERVENTIONS:
Drug: Tarceva — Tarceva (erlotinib hydrochloride) given alone, at 150 mg by mouth daily.
  Other Names: Erlotinib hydrochloride; OSI-774

SUMMARY:
The goal of this clinical research study is to learn if Tarceva® (erlotinib hydrochloride) can help control triple receptor-negative breast cancer. The safety of this drug will also be studied.

Objectives:

To assess the clinical efficacy, biologic effects and safety of the EGFR inhibitor erlotinib in the treatment of patients with 'triple receptor-negative' metastatic carcinoma of the breast.

Primary endpoints:

1) Time to progression (TTP)

Secondary endpoints:

1. clinical benefit rate as defined by complete and partial response and stable disease
2. overall survival (OS)
3. safety profile and tolerability of erlotinib
4. biologic correlative studies

DETAILED DESCRIPTION:
The Study Drug:

Erlotinib hydrochloride is designed to block the activity of a protein found on the surface of many tumor cells that may control tumor growth and survival. This may stop tumors from growing.

Screening Tests:

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study.

* Blood (about 5 teaspoons) will be drawn for routine tests.
* If you have had a biopsy at M. D. Anderson, your leftover tissue will be used to confirm the breast cancer is triple receptor-negative.
* If you have had a biopsy at another location, a part of that biopsy will be collected and tested to make sure that the breast cancer is triple receptor-negative.
* You will have imaging scans, such as computed tomography (CT) or bone scans, to check the status of the disease.
* If no tissue is available to check the status of the disease, you will have a breast biopsy. To collect a tumor biopsy, the affected area is numbed with anesthetic, and a small amount of tissue is withdrawn through a large needle.

Study Drug Dose Level:

If you are found to be eligible to take part in this study, you will take erlotinib hydrochloride by mouth once a day, every day, between breakfast and lunch. You should take erlotinib hydrochloride 1 hour before or 2 hours after eating. It should be taken at the same time each day.

Study Visits:

Every 8 weeks, the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 5 teaspoons) will be drawn for routine tests.
* You will have the same imaging scans that were performed at screening to check the status of the disease.
* You will be asked about any side effects you may be experiencing.

Length of Study:

You may remain on this study for as long as you are benefiting. You will be taken off this study if the disease gets worse or intolerable side effects occur.

End-of-Study Visit:

You will have an end-of-study visit once you are off this study. The following tests and procedures will be performed at this visit.

Blood (about 5 teaspoons) will be drawn for routine tests. You will have the same imaging scans repeated to check the status of the disease.

This is an investigational study. Erlotinib hydrochloride is FDA approved and commercially available for the treatment of advanced lung cancer and advanced pancreatic cancer. Its use in breast cancer is investigational. Up to 50 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologic confirmation of metastatic (stage IV) 'triple receptor-negative' breast cancer. Tissue must be available at baseline or agree to biopsy. The diagnosis of 'triple receptor-negative' breast cancer requires that either the primary tumor or a metastatic deposit be shown to be negative for estrogen receptors (ER) and progesterone receptors (PR) by immunohistochemistry (IHC) and for HER2/neu by IHC (i.e. a score of 0 and 1+) or fluorescent in situ hybridization (FISH).
2. EGFR protein expression and gene copy number will be evaluated on stored tissue sample at a later time. Unstained slides, a block, or agreement for biopsy is required for study participation.
3. Patients with metastatic breast cancer to any distant site are eligible once their disease is clinically/radiologically measurable
4. Patients must have disease which is resistant to taxanes and anthracyclines. There is no limit to the number of previous therapies for metastatic disease.
5. Patients are eligible if they have not had prior exposure to an EGFR inhibitor (e.g.Gefitinib, Erlotinib) or antibody (e.g. Cetuximab).
6. Availability of tissue blocks and/or fresh/frozen tumor samples is an eligibility requirement in order to run the EGFR IHC, FISH and to confirm, if needed ER, PR and HER2/neu status.
7. Patients may, but are not required, to have a repeat tumor biopsy performed on study entry prior to beginning therapy and also early during study therapy for correlative studies.
8. Patients with 'triple receptor-negative' metaplastic breast cancers are eligible if they meet the criterion of EGFR overexpression.
9. Patients must sign an informed consent indicating that they are aware of the investigational nature of the study, in keeping with institutional policy
10. Patients must have tissue blocks available from previous primary tumor surgery or biopsy or from a previous biopsy of metastatic disease for EGFR status assessment and for correlative studies
11. Patients should have adequate bone marrow function, as defined by peripheral granulocyte count of >/= 1500/mm^3, and a platelet count >/= 100000/ mm^3. Patients must have adequate liver function with a bilirubin within 1.5 times the upper limit of normal (ULN). Transaminases (SGPT) may be up to 5 * the ULN and alkaline phosphatase may be up to 5 * ULN
12. Patients should have adequate renal function (serum creatinine </= 1.5 times the ULN)
13. Negative pregnancy test for a woman of childbearing potential
14. Women of childbearing potential must use a reliable and appropriate contraceptive method during the study
15. Patients with a performance status of 2 or better by World Health Organization (W.H.O.)

Exclusion Criteria:

1. Patients with uncompensated congestive cardiac failure are not eligible
2. Patients with a myocardial infarction in the previous 12 months are not eligible
3. Patients with central nervous system (CNS) metastases are not eligible
4. Patients with an organ allograft
5. Patients with a serious concurrent infection or illness including, but not limited to, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness that would limit compliance with study requirements

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Hennessy, MD/Asst Prof, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: July 22, 2008 to November 03, 2010. All recruitment done at UT MD Anderson Cancer Center.
Pre-assignment Details: Study terminated early due to slow accrual. Eleven patients were enrolled, only three received treatment.
Period: Overall Study
Arm/Group | Tarceva Daily
Started | 11
Completed | 3
Not Completed | 8
Not completed — Screen failures | 8

BASELINE CHARACTERISTICS:
Arm/Group | Tarceva Daily
Number analyzed (Participants) | 11
Age Continuous [Mean (Full Range); unit: years] | 52 [37 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP)
Description: Time to progression calculated from the date of study entry to the date of disease progression or death. Progression of disease is defined by RECIST (Response Evaluation Criteria In Solid Tumors) criteria, as measurable increase in the smallest dimension of any target or not-target lesion, or the appearance of new lesions, since baseline. Confirmed response based on two tumor assessments (imaging) separated by at least 4 weeks.
Time Frame: Baseline to disease progression, up to 22 months with follow up.
Population: Study terminated early, unable to complete overall analysis due to insufficient data.
Measure: Number; unit: months
Arm/Group | Tarceva Daily
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 16 months
Description: Only 3 of 11 participants received treatment, therefore Adverse Events were only collected on those 3 participants.
Arm/Group | Tarceva Daily
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tarceva Daily (N=3)
Diarrhea (Gastrointestinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tarceva Daily (N=3)
Alanine aminotransferase (Blood and lymphatic system disorders) | 3
Aspartate aminotransferase increased (Investigations) | 2
Alkaline phosphotase increased (Investigations) | 1
Hemoglobin decreased (Blood and lymphatic system disorders) | 1
Serum magnesium decreased (Investigations) | 1
Serum sodium decreased (Investigations) | 1
Lymphopenia (Blood and lymphatic system disorders) | 2
Dermatology/Skin (Other) - skin rash (Skin and subcutaneous tissue disorders) | 3
Stomatitis (Metabolism and nutrition disorders) | 3
Diarrhea (Gastrointestinal disorders) | 3
Metabolic/Laboratory (Other) - carbon dioxide (Metabolism and nutrition disorders) | 1
Ocular/Visual (Other) - red eyes (Eye disorders) | 2
Fatigue (General disorders) | 2
Localized edema (General disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Hand-and-foot syndrome (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 1
Musculoskeletal (other) - leg cramping (Musculoskeletal and connective tissue disorders) | 1
Pulmonary (other) - sore in nostril (Respiratory, thoracic and mediastinal disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No